CLINICAL TRIAL: NCT02052245
Title: Longitudinal Composition of Human Milk for Term and Preterm Infants
Brief Title: Pre/Term Milk Profiling
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 11.39.NRC
Record Dates: First submitted 2013-10-08; First posted 2014-02-03 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Preterm Milk; Term Milk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subject delivering preterm baby
- Subject delivering term baby

SUMMARY:
This study aims for an in-depth characterization of human milk of mothers who delivered prematurely to decipher differences with milk of mothers who delivered at the expected term, with a particular focus on milk proteins

ELIGIBILITY:
Inclusion Criteria:

* Having obtained informed consent
* Group 1 (term delivery): Gestational age between 37 0/7 and not above 41 6/7 weeks
* Group 2 (preterm delivery): Gestational age between 28 0/7 and 32 6/7 weeks
* Age: Mother ≥ 18 years old
* Partial or total breast feeding
* Having a freezer compartment at home (approx. -18°C)
* Good understanding of the French language

Exclusion Criteria:

* Suffering from diabetes (type I or II) before pregnancy
* Alcohol consumption: more than 1 standard drink / day
* Drug addicted
* Subject who cannot be expected to comply with the study procedures.
* Currently participating in an interventional therapeutic clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mothers who will breast feed their baby
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Quantification of total protein concentration in human milk | from delivery, up to 4 months

SECONDARY OUTCOMES:
Quantification of total lipids and carbohydrates | From delivery, up to 4 months
Determination of Calcium and Phosphorous content | From delivery, up to 4 months
Determination of peptide profiles and content | From delivery, up to 4 months
Determination of miRNA content | From delivery, up to 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of neonatology - Avenue Pierre Decker 2, Lausanne, Switzerland

REFERENCES:
- [Derived] Garcia-Rodenas CL, De Castro CA, Jenni R, Thakkar SK, Beauport L, Tolsa JF, Fischer-Fumeaux CJ, Affolter M. Temporal changes of major protein concentrations in preterm and term human milk. A prospective cohort study. Clin Nutr. 2019 Aug;38(4):1844-1852. doi: 10.1016/j.clnu.2018.07.016. Epub 2018 Jul 26. PMID 30093147